CLINICAL TRIAL: NCT01577836
Title: Medico-economic Comparison of Robot-assisted Radical Prostatectomy Using the da Vinci System Versus Radical Prostatectomy Via Laparotomy
Brief Title: Medico-economic Comparison of Robot-assisted Radical Prostatectomy Versus Radical Prostatectomy Via Laparotomy
Acronym: RoboProstate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOI/2011/SD-03; 2011-A01385-36 (Other: ANSM)
Record Dates: First submitted 2012-04-13; First posted 2012-04-16 (Estimated); Last update posted 2025-12-12 (Actual); Status verified 2023-06

CONDITIONS: Prostatic Neoplasms
Keywords: Radical prostatectomie; Robotic assistance; Laparotomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Robotic assistance, Nîmes (Experimental): The patients in this group will undergo robot-assisted radical prostatectomy at the University Hospital of Nîmes.
  Interventions: Procedure: Robot-assisted radical prostatectomy
- Laparotomy, Marseilles (Active Comparator): The patients in this group will undergo radical prostatectomy via traditional laparotomy at the University Hospital Marseillles.
  Interventions: Procedure: Radical prostatectomy via laparotomy

INTERVENTIONS:
Procedure: Robot-assisted radical prostatectomy — Transperitoneal robot-assisted radical prostatectomy technique with the Da Vinci S
  Arms: Robotic assistance, Nîmes
Procedure: Radical prostatectomy via laparotomy — Classic radical prostatectomy via open retropubic approach
  Arms: Laparotomy, Marseilles

SUMMARY:
The main objective of the study is to estimate and compare the overall cost of care of patients over 60 months of follow-up between two groups: (1) patients undergoing robot-assisted radical prostatectomy using the Da Vinci system versus (2) patients undergoing robot-assisted radical prostatectomy via laparotomy.

The time horizon of the main objective changes to 60 months (due to the opportunity to access patient care consumption from the National Health Data System).

DETAILED DESCRIPTION:
The secondary objectives of this research are to compare the following between the two groups:

* The actual cost of the surgical prostatectomy.
* Erectile function at 0, 1, 6, 12 and 24
* Oncological results at 1, 6, 12 and 24 months.
* Functional results at 0, 1, 6, 12 and 24 months.
* Quality of life at 0, 1, 6, 12 and 24 months.
* Complication rates at 1 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 24 months of follow up
* Patient has localised prostate cancer
* Patient is eligible for radical prostatectomy

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* Patient has a contraindication for a treatment necessary for this study
* Patients with psychiatric disorders

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-11-26 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
Overall cost (€) of patient care | 60 months
  Cost of surgical treatment of localized prostate cancer by radical prostatectomy (robot-assisted or conventional retropubic laparotomy) and its follow-up for 5 years. All medical resources consumed will be evaluated during the first 5 years after surgery.

SECONDARY OUTCOMES:
Cost (€) of surgery via micro-costing | Day 1
  All human and material resources necessary for carrying out a prostatectomy will be evaluated.
Change in erectile function | baseline to 1 month
  the International Index of Erectile Function (IIEF-15) will be used.
Change in erectile function | baseline to 6 months
  the International Index of Erectile Function (IIEF-15) will be used.
Change in erectile function | baseline to 12 months
  the International Index of Erectile Function (IIEF-15) will be used.
Change in erectile function | baseline to 24 months
  the International Index of Erectile Function (IIEF-15) will be used.
the % of positive margins after resection | baseline (Day 1)
presence/absence of PSA (Prostate Specific Antigen ) > 0.2 ng/ml (recurrence) | 1 month
presence/absence of PSA (Prostate Specific Antigen ) > 0.2 ng/ml (recurrence) | 6 months
presence/absence of PSA (Prostate Specific Antigen ) > 0.2 ng/ml (recurrence) | 12 months
presence/absence of PSA (Prostate Specific Antigen ) > 0.2 ng/ml (recurrence) | 24 months
Change in function as estimated by the PR25 questionnaire | baseline to 1 month
Change in function as estimated by the PR25 questionnaire | baseline to 6 months
Change in function as estimated by the PR25 questionnaire | baseline to 12 months
Change in function as estimated by the PR25 questionnaire | baseline to 24 months
Change in quality of life as estimated by the QLQC-30 questionnaire | baseline to 1 month
Change in quality of life as estimated by the QLQC-30 questionnaire | baseline to 6 months
Change in quality of life as estimated by the QLQC-30 questionnaire | baseline to 12 months
Change in quality of life as estimated by the QLQC-30 questionnaire | baseline to 24 months
Presence/absence of complications (Clavien) | 1 month
  The Clavien classification will be used (Clavien, P.A., Sanabria J.R., et S.M. Strasberg. 1992. Proposed classification of complications of surgery with examples of utility in cholecystectomy. Suregry 111 (5): 518-526.)
Presence/absence of complications (Clavien) | 24 months
  The Clavien classification will be used (Clavien, P.A., Sanabria J.R., et S.M. Strasberg. 1992. Proposed classification of complications of surgery with examples of utility in cholecystectomy. Suregry 111 (5): 518-526.)
Presence/absence of complications (Pentafecta) | 1 month
  The Pentafecta classification will be used.
Presence/absence of complications (Pentafecta) | 24 months
  The Pentafecta classification will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Droupy, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (3):
- France (3):
  - APHM - Hôpital de la Conception, Marseille
  - Clinique Beau Soleil, Montpellier
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes

REFERENCES:
- [Result] Bouvet S, Chkair S, Daures JP, Kabani S; OptiPRobot Study Group; Chevallier T, Lechevallier E, Droupy S. Robot-assisted approach versus open surgery and conventional laparoscopy for radical prostatectomy for prostate cancer: a micro-costing study. Health Econ Rev. 2025 Jul 5;15(1):55. doi: 10.1186/s13561-025-00652-5. PMID 40616606